CLINICAL TRIAL: NCT00564304
Title: Nasal Potential Difference Measurement in Infants
Brief Title: NPD Measurement in Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: will004-HMO-CTIL
Record Dates: First submitted 2007-11-25; First posted 2007-11-27 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Cystic Fibrosis
Keywords: Nasal Potential Difference
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Nasal Potential Difference measurements (NPD) have been performed in Israel since 1996. NPD measurements are used to assess the voltage across nasal epithelium, which correlates with the transport of sodium and chloride across cell membranes. NPD was first demonstrated to be abnormal in Cystic Fibrosis (CF) in 1981 and the technique has since been used to increase our understanding of this condition. It is now established as an important diagnostic tool and more recently has been used to assess the effectiveness of new treatments such as gene and alternative therapy (Knowles 1995; Wilschanski 2003).

The nasal cavity is accessible which makes it a good site to examine the ion transport characteristics of airway epithelia. Less than a centimetre into the nose the squamous ("skin type") epithelium becomes ciliated pseudocolumnar epithelium, characteristic of the proximal airways.

The change in NPD with the perfusion of different solutions is demonstrated. By employing NPD protocols with perfusion of different solutions and drugs, different aspects of the nasal ion transport characteristics can be examined. In CF, this ion transport profile is abnormal and the NPD measurement has a number of features that differentiate CF from non-CF. This methodology is well established for measurements in subjects over 6 years of age.

Measurements on smaller children and infants have been very difficult to perform. We propose a new method using smaller, single lumen catheters with much lower perfusion rates (0.2 ml/min compared to up to 5 ml/min with the adult method) .Perfusion measurements will be possible in newly born infants. Obviously this opens up the potential for using NPD as a diagnostic test in babies. This is important as the diagnosis of CF is often difficult to make or refute in babies because of the problems in collecting enough sweat. This may be the ideal diagnostic test for CF in the neonatal nursery in infants with meconium plug syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age below 6 years
* Patients who suspected for CF due to pulmonary and/or gastrointestinal symptoms

Exclusion Criteria:

* Age over 6 years

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children below age of 6 years who suspected for Cystic Fibrosis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Study Completion 2010-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wilschanski, Dr., Principal Investigator — Hadassah Medical Organization